CLINICAL TRIAL: NCT03777774
Title: Vacuum Drains vs Passive Drains vs no Drains in Decompressive Craniectomies - A Randomized Controlled Trial on Subgaleal Drain Complication Rates
Brief Title: Subgaleal Drains in Decompressive Craniectomies
Acronym: VADER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Sam Jo Ee, Principal investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VADER 1.0
Record Dates: First submitted 2018-12-11; First posted 2018-12-17 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Hematoma Intracranial; Hydrocephalus; Surgical Site Infection; Wound Breakdown; Bradycardia; Hypotension Postprocedural
Keywords: Decompressive craniectomy; subgaleal drain; subgaleal hematoma; Post craniectomy hydrocephalus; surgical site infection; Bradycardia; Hypotension; Wound breakdown
MeSH Terms: conditions — Hydrocephalus; Surgical Wound Infection; Surgical Wound Dehiscence; Bradycardia; Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Patients will be randomized only after the closing stage of decompressive craniectomy to avoid surgeon bias
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No subgaleal drains (Active Comparator): Drains will be placed during closing stage of craniectomy but will be clamped so that no drainage takes place. Drains can be opened if needed
  Interventions: Procedure: No Redon subgaleal drains
- Passive subgaleal drains (Active Comparator): Passive non-vacuum drains will be placed during closing stage of craniectomy
  Interventions: Procedure: Passive Redon subgaleal drains
- Vacuum subgaleal drains (Active Comparator): Active vacuum drains will be placed during closing stage of craniectomy
  Interventions: Procedure: Vacuum Redon subgaleal drains

INTERVENTIONS:
Procedure: Passive Redon subgaleal drains — Passive non-vacuum subgaleal drains will be placed during closing stage of craniectomy. Drain used is closed suction drain system (3.2 mm in outer diameter, 10 French, round and transparent polyvinyl chloride tube with a 400 mL Redon bottle spring evacuator chamber; Privac, Primed, Germany)
  Other Names: Non-vacuum drain
  Arms: Passive subgaleal drains
Procedure: Vacuum Redon subgaleal drains — Active vacuum subgaleal drains will be placed during the closing stage of craniectomy. Drain used is closed suction drain system (3.2 mm in outer diameter, 10 French, round and transparent polyvinyl chloride tube with a 400 mL Redon bottle spring evacuator chamber; Privac, Primed, Germany)
  Other Names: Active drains
  Arms: Vacuum subgaleal drains
Procedure: No Redon subgaleal drains — A subgaleal drain will be placed during the closing stage of craniectomy but it will be clamped. The drain will be unclamped if necessary. Drain used is closed suction drain system (3.2 mm in outer diameter, 10 French, round and transparent polyvinyl chloride tube with a 400 mL Redon bottle spring evacuator chamber; Privac, Primed, Germany)
  Other Names: no drains
  Arms: No subgaleal drains

SUMMARY:
This research is about the use of subgaleal drains to prevent accumulation of blood under the skin in patients undergoing surgery to remove part of the skull(craniectomy) and its associated complications. There have been early research that shows usage of subgaleal drains maybe related to increase in complication rates after craniectomy. These complications include hydrocephalus (accumulation of fluid in the brain), new hemorrhages, infection and low blood pressure. The investigators are performing this research to determine which type of subgaleal drains would produce the least complications. With this knowledge, the investigators would be able to reduce the amount of complications for future patients that undergo surgery to remove part of the skull.

The purpose of this study is to determine the rate of complications in the 3 different groups of patients using the different types of drains under the skin in surgeries that involve removal of part of the skull.

All participants will undergo the required surgery to remove part of the skull (craniectomy). Participants will then be randomly assigned to either one of 3 groups which are the vacuum drain group, passive drain group or no drain group.Participants in the vacuum drain group will have vacuum drains inserted during the closing stage of the surgery. Participants in the passive drain group will have passive drains inserted during the closing stage of the surgery. Participants in the no drain group will have a drain inserted during the closing stage of the procedure but the drain will remained closed.

Data will then be collected and analysed to determine if the type of drains influence the rate of complications in craniectomy

DETAILED DESCRIPTION:
Prophylactic subcutaneous drains in surgery have generally been used for detection and drainage of hematomas or excessive secretions. In the past three decades, multiple surgical disciplines have conducted studies to determine the necessity of vacuum drains or even the need of drains altogether and a meta-analysis found that many operations can be carried out safely without prophylactic drainage.

In addition to that, drains have been associated with complications. A few of them include wound infections, injury to tissues, source of discomfort and pain during removal, limiting mobility and additional scarring.

Of all the cranial surgeries, the most commonly performed surgery is decompressive craniectomy. This surgery has been an increasingly common surgical procedure for the neurosurgical community as there is clear evidence from numerous studies that support decompressive craniectomy as a life-saving surgical procedure in traumatic brain injury, malignant middle cerebral artery infarction and spontaneous intracerebral haemorrhage.

Decompressive craniectomies have been associated with many complications including subdural effusions (49%), post-craniectomy hydrocephalus (14%), subgaleal hematomas and new remote hematomas (10.2%). These complications may just be due to the surgery itself. But it may still be possible that these complications are worsened or arise solely due to the routine use of the vacuum drain.

As the utility of decompressive craniectomy increases, efforts should be made to reduce the complications related to it. Studies have been done to optimize and standardize the technique of decompressive craniectomy but the necessity to use the vacuum drains and the possible contribution that these drains may have to the complications of decompressive craniectomies have been overlooked so far. There have been no randomized studies to compare usage of subgaleal vacuum drains, subgaleal passive drains and the omission of subgaleal drains in neurosurgical practice to date.

Usage of subgaleal vacuum drains for decompressive craniectomies have been the usual practice so far to prevent subgaleal hematoma collection. However, this practice is not backed by any strong evidence that these vacuum drains actually deter subgaleal hematoma collection. On top of that, these vacuum drains may itself be causing complications that have not been discovered before. The usual complications associated with prophylactic vacuum drains are surgical site infections and wound breakdown. There are other complications that could be attributed to the routine usage of prophylactic vacuum drains. These include new remote intracranial hematomas, post craniectomy hydrocephalus and bradycardia or hypotension during the skin closure stage of craniectomy.

The investigators plan to compare the complication rates of vacuum drains, passive drains and no drains in decompressive craniectomy. These 3 groups include a group with active vacuum drains, another group with passive non-vacuum drains and a group without any drains. The current practice is to use active or passive vacuum drains as prophylactic drains in patients undergoing decompressive craniectomy.

The complication rates to be studied are:

1. subgaleal hematoma thickness
2. new remote hematomas,
3. post craniectomy hydrocephalus,
4. surgical site infection,
5. wound breakdown,
6. bradycardia/hypotension during closing stage of craniectomy
7. and functional outcomes of patients at 6 months

If the rates of complications in the groups without a drain or a passive drain are lower or equal to that of the group with active drains, this study may change the paradigm of prophylactic drain usage in decompressive craniectomies

ELIGIBILITY:
Inclusion Criteria:

* patients with indication for decompressive craniectomy as decided by the neurosurgeon in-charge. Indications maybe for traumatic intracranial bleed, spontaneous intracranial bleed and malignant middle cerebral artery territory infarction
* Written informed consent by legal representative of patient

Exclusion Criteria:

* history of recent antiplatelet or anticoagulant use
* patients with evidence of coagulopathy or thrombocytopenia from lab results
* possible disseminated intravascular coagulation preoperatively
* Presence of hydrocephalus preoperatively

Ages: 0 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Subgaleal hematomas | 24 hours +/- 12 hours post craniectomy
  Mean maximum thickness and volume of subgaleal hematomas as post craniectomy complication. Defined as maximum thickness and volume (using XYZ/2 formula) of subgaleal hematoma on CT brain post craniectomy.

SECONDARY OUTCOMES:
New remote hematomas | 1 week post craniectomy
  Rate of new remote hematomas. Defined as hematomas not previously seen on earlier CT brains but seen on post operative CT brain that cannot be explained by direct connection or complication from the original hematomas
Surgical site infection | 1 month post craniectomy
  Rate of surgical site infection. Defined as purulent or serous discharge from the surgical site with clinical signs of inflammation
Wound breakdown | 1 month post craniectomy
  Rate of wound breakdown. Defined as spontaneous separation of sutured edges
Bradycardia or hypotension during skin closure stage. | end of surgery till 30 minutes after surgery has ended
  Rate of bradycardia or hypotension during skin closure stage. Bradycardia defined as <60 beat per minute, hypotension defined as BP <90/60 mmHg, that cannot be clearly explained by other possible causes
Post craniectomy hydrocephalus | 6 months post craniectomy
  Rate of post craniectomy hydrocephalus. Defined as radiographic and clinical evidence of hydrocephalus post craniectomy
Functional outcome | 6 months post craniectomy
  Modified Rankin Scale(MRS) score on 6 months post craniectomy
  MRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities
  The scale runs from 0-6, running from perfect health without symptoms to death.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

CONTACTS AND LOCATIONS:
Overall Officials: Jo Ee Sam, Principal Investigator — Hospital University Sains Malaysia
Locations (2):
- Malaysia (2):
  - Hospital University Sains Malaysia, Kubang Kerian, Kelantan
  - Sarawak General Hospital, Kuching, Sarawak

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kosins AM, Scholz T, Cetinkaya M, Evans GRD. Evidence-based value of subcutaneous surgical wound drainage: the largest systematic review and meta-analysis. Plast Reconstr Surg. 2013 Aug;132(2):443-450. doi: 10.1097/PRS.0b013e3182958945. PMID 23584625
- [Background] Cruse PJ, Foord R. A five-year prospective study of 23,649 surgical wounds. Arch Surg. 1973 Aug;107(2):206-10. doi: 10.1001/archsurg.1973.01350200078018. No abstract available. PMID 4719566
- [Background] Nalbach SV, Ropper AE, Dunn IF, Gormley WB. Craniectomy-associated Progressive Extra-Axial Collections with Treated Hydrocephalus (CAPECTH): redefining a common complication of decompressive craniectomy. J Clin Neurosci. 2012 Sep;19(9):1222-7. doi: 10.1016/j.jocn.2012.01.016. Epub 2012 Jun 20. PMID 22727206
- [Background] Vedantam A, Yamal JM, Hwang H, Robertson CS, Gopinath SP. Factors associated with shunt-dependent hydrocephalus after decompressive craniectomy for traumatic brain injury. J Neurosurg. 2018 May;128(5):1547-1552. doi: 10.3171/2017.1.JNS162721. Epub 2017 Jun 16. PMID 28621627
- [Background] Manfiotto M, Mottolese C, Szathmari A, Beuriat PA, Klein O, Vinchon M, Gimbert E, Roujeau T, Scavarda D, Zerah M, Di Rocco F. Decompressive craniectomy and CSF disorders in children. Childs Nerv Syst. 2017 Oct;33(10):1751-1757. doi: 10.1007/s00381-017-3542-7. Epub 2017 Sep 6. PMID 29149390
- [Background] Weintraub AH, Gerber DJ, Kowalski RG. Posttraumatic Hydrocephalus as a Confounding Influence on Brain Injury Rehabilitation: Incidence, Clinical Characteristics, and Outcomes. Arch Phys Med Rehabil. 2017 Feb;98(2):312-319. doi: 10.1016/j.apmr.2016.08.478. Epub 2016 Sep 23. PMID 27670926
- [Background] Powers AK, Neal MT, Argenta LC, Wilson JA, DeFranzo AJ, Tatter SB. Vacuum-assisted closure for complex cranial wounds involving the loss of dura mater. J Neurosurg. 2013 Feb;118(2):302-8. doi: 10.3171/2012.10.JNS112241. Epub 2012 Nov 16. PMID 23157181
- [Background] Wilkie KP, Nagra G, Johnston M. A MATHEMATICAL ANALYSIS OF PHYSIOLOGICAL AND MOLECULAR MECHANISMS THAT MODULATE PRESSURE GRADIENTS AND FACILITATE VENTRICULAR EXPANSION IN HYDROCEPHALUS. Int J Numer Anal Model B. 2012;316:65-81. PMID 25678938
- [Background] Waziri A, Fusco D, Mayer SA, McKhann GM 2nd, Connolly ES Jr. Postoperative hydrocephalus in patients undergoing decompressive hemicraniectomy for ischemic or hemorrhagic stroke. Neurosurgery. 2007 Sep;61(3):489-93; discussion 493-4. doi: 10.1227/01.NEU.0000290894.85072.37. PMID 17881960
- [Background] Yadav YR, Parihar V, Chourasia ID, Bajaj J, Namdev H. The role of subgaleal suction drain placement in chronic subdural hematoma evacuation. Asian J Neurosurg. 2016 Jul-Sep;11(3):214-8. doi: 10.4103/1793-5482.145096. PMID 27366247
- [Background] Van Roost D, Thees C, Brenke C, Oppel F, Winkler PA, Schramm J. Pseudohypoxic brain swelling: a newly defined complication after uneventful brain surgery, probably related to suction drainage. Neurosurgery. 2003 Dec;53(6):1315-26; discussion 1326-7. doi: 10.1227/01.neu.0000093498.08913.9e. PMID 14633298
- [Background] Huang YH, Lee TC, Lee TH, Yang KY, Liao CC. Remote epidural hemorrhage after unilateral decompressive hemicraniectomy in brain-injured patients. J Neurotrauma. 2013 Jan 15;30(2):96-101. doi: 10.1089/neu.2012.2563. PMID 23013227
- [Background] Meguro T, Terada K, Hirotsune N, Nishino S, Asano T. Postoperative extradural hematoma after removal of a subgaleal drainage catheter--case report. Neurol Med Chir (Tokyo). 2007 Jul;47(7):314-6. doi: 10.2176/nmc.47.314. PMID 17652918
- [Background] Kurland DB, Khaladj-Ghom A, Stokum JA, Carusillo B, Karimy JK, Gerzanich V, Sahuquillo J, Simard JM. Complications Associated with Decompressive Craniectomy: A Systematic Review. Neurocrit Care. 2015 Oct;23(2):292-304. doi: 10.1007/s12028-015-0144-7. PMID 26032808
- [Background] Chang V, Hartzfeld P, Langlois M, Mahmood A, Seyfried D. Outcomes of cranial repair after craniectomy. J Neurosurg. 2010 May;112(5):1120-4. doi: 10.3171/2009.6.JNS09133. PMID 19612971
- [Background] Sobani ZA, Shamim MS, Zafar SN, Qadeer M, Bilal N, Murtaza SG, Enam SA, Bari ME. Cranioplasty after decompressive craniectomy: An institutional audit and analysis of factors related to complications. Surg Neurol Int. 2011;2:123. doi: 10.4103/2152-7806.85055. Epub 2011 Sep 17. PMID 22059118
- [Background] Choi SY, Yoon SM, Yoo CJ, Park CW, Kim YB, Kim WK. Necessity of Surgical Site Closed Suction Drain for Pterional Craniotomy. J Cerebrovasc Endovasc Neurosurg. 2015 Sep;17(3):194-202. doi: 10.7461/jcen.2015.17.3.194. Epub 2015 Sep 30. PMID 26523255
- [Background] Guangming Z, Huancong Z, Wenjing Z, Guoqiang C, Xiaosong W. Should epidural drain be recommended after supratentorial craniotomy for epileptic patients? Surg Neurol. 2009 Aug;72(2):138-41; discussion 141. doi: 10.1016/j.surneu.2008.06.014. PMID 19608006
- [Background] Shi SS, Zhang GL, Zeng T, Lin YF. Posttraumatic hydrocephalus associated with decompressive cranial defect in severe brain-injured patients. Chin J Traumatol. 2011;14(6):343-7. PMID 22152137
- [Background] Meyerson JM. A Brief History of Two Common Surgical Drains. Ann Plast Surg. 2016 Jan;77(1):4-5. doi: 10.1097/SAP.0000000000000734. PMID 26808754
- [Background] Morris AM. A controlled trial of closed wound suction. Br J Surg. 1973 May;60(5):357-9. doi: 10.1002/bjs.1800600509. No abstract available. PMID 4574786
- [Background] Hutchinson PJ, Kolias AG, Timofeev IS, Corteen EA, Czosnyka M, Timothy J, Anderson I, Bulters DO, Belli A, Eynon CA, Wadley J, Mendelow AD, Mitchell PM, Wilson MH, Critchley G, Sahuquillo J, Unterberg A, Servadei F, Teasdale GM, Pickard JD, Menon DK, Murray GD, Kirkpatrick PJ; RESCUEicp Trial Collaborators. Trial of Decompressive Craniectomy for Traumatic Intracranial Hypertension. N Engl J Med. 2016 Sep 22;375(12):1119-30. doi: 10.1056/NEJMoa1605215. Epub 2016 Sep 7. PMID 27602507
- [Background] Alexander P, Heels-Ansdell D, Siemieniuk R, Bhatnagar N, Chang Y, Fei Y, Zhang Y, McLeod S, Prasad K, Guyatt G. Hemicraniectomy versus medical treatment with large MCA infarct: a review and meta-analysis. BMJ Open. 2016 Nov 24;6(11):e014390. doi: 10.1136/bmjopen-2016-014390. PMID 27884858
- [Background] Hemphill JC 3rd, Greenberg SM, Anderson CS, Becker K, Bendok BR, Cushman M, Fung GL, Goldstein JN, Macdonald RL, Mitchell PH, Scott PA, Selim MH, Woo D; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology. Guidelines for the Management of Spontaneous Intracerebral Hemorrhage: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Jul;46(7):2032-60. doi: 10.1161/STR.0000000000000069. Epub 2015 May 28. PMID 26022637
- [Background] Honeybul S, Ho KM. Long-term complications of decompressive craniectomy for head injury. J Neurotrauma. 2011 Jun;28(6):929-35. doi: 10.1089/neu.2010.1612. Epub 2011 Jun 1. PMID 21091342
- [Background] Ding J, Guo Y, Tian H. The influence of decompressive craniectomy on the development of hydrocephalus: a review. Arq Neuropsiquiatr. 2014 Sep;72(9):715-20. doi: 10.1590/0004-282x20140106. PMID 25252237
- [Background] Rahme R, Weil AG, Sabbagh M, Moumdjian R, Bouthillier A, Bojanowski MW. Decompressive craniectomy is not an independent risk factor for communicating hydrocephalus in patients with increased intracranial pressure. Neurosurgery. 2010 Sep;67(3):675-8; discussion 678. doi: 10.1227/01.NEU.0000383142.10103.0B. PMID 20651634
- [Background] Zhou L, Yu J, Sun L, Han Y, Wang G. Overdrainage after ventriculoperitoneal shunting in a patient with a wide depressed skull bone defect: The effect of atmospheric pressure gradient. Int J Surg Case Rep. 2016;29:11-15. doi: 10.1016/j.ijscr.2016.10.012. Epub 2016 Oct 15. PMID 27810603
- [Background] De Bonis P, Pompucci A, Mangiola A, Rigante L, Anile C. Post-traumatic hydrocephalus after decompressive craniectomy: an underestimated risk factor. J Neurotrauma. 2010 Nov;27(11):1965-70. doi: 10.1089/neu.2010.1425. PMID 20812777
- [Background] Anile C, De Bonis P, Di Chirico A, Ficola A, Mangiola A, Petrella G. Cerebral blood flow autoregulation during intracranial hypertension: a simple, purely hydraulic mechanism? Childs Nerv Syst. 2009 Mar;25(3):325-35; discussion 337-40. doi: 10.1007/s00381-008-0749-7. Epub 2009 Jan 17. PMID 19152096
- [Background] Takeuchi S, Nawashiro H, Wada K, Takasato Y, Masaoka H, Hayakawa T, Nagatani K, Otani N, Osada H, Shima K. Ventriculomegaly after decompressive craniectomy with hematoma evacuation for large hemispheric hypertensive intracerebral hemorrhage. Clin Neurol Neurosurg. 2013 Mar;115(3):317-22. doi: 10.1016/j.clineuro.2012.05.026. Epub 2012 Jun 21. PMID 22727212
- [Background] Jiao QF, Liu Z, Li S, Zhou LX, Li SZ, Tian W, You C. Influencing factors for posttraumatic hydrocephalus in patients suffering from severe traumatic brain injuries. Chin J Traumatol. 2007 Jun;10(3):159-62. PMID 17535639
- [Background] Honeybul S, Ho KM. Incidence and risk factors for post-traumatic hydrocephalus following decompressive craniectomy for intractable intracranial hypertension and evacuation of mass lesions. J Neurotrauma. 2012 Jul 1;29(10):1872-8. doi: 10.1089/neu.2012.2356. PMID 22583391
- [Background] Pandey S, Jin Y, Gao L, Zhou CC, Cui DM. Negative-Pressure Hydrocephalus: A Case Report on Successful Treatment Under Intracranial Pressure Monitoring with Bilateral Ventriculoperitoneal Shunts. World Neurosurg. 2017 Mar;99:812.e7-812.e12. doi: 10.1016/j.wneu.2016.12.049. Epub 2016 Dec 23. PMID 28017745
- [Background] Yadav M, Nikhar SA, Kulkarni DK, Gopinath R. Cardiac Arrest after Connecting Negative Pressure to the Subgaleal Drain during Craniotomy Closure. Case Rep Anesthesiol. 2014;2014:146870. doi: 10.1155/2014/146870. Epub 2014 May 22. PMID 24963414
- [Background] Quinn TM, Taylor JJ, Magarik JA, Vought E, Kindy MS, Ellegala DB. Decompressive craniectomy: technical note. Acta Neurol Scand. 2011 Apr;123(4):239-44. doi: 10.1111/j.1600-0404.2010.01397.x. PMID 20637010
- [Background] Huang X, Wen L. Technical considerations in decompressive craniectomy in the treatment of traumatic brain injury. Int J Med Sci. 2010 Nov 8;7(6):385-90. doi: 10.7150/ijms.7.385. PMID 21103073
- [Background] Roth J, Galeano E, Milla S, Hartmannsgruber MW, Weiner HL. Multiple epidural hematomas and hemodynamic collapse caused by a subgaleal drain and suction-induced intracranial hypotension: case report. Neurosurgery. 2011 Jan;68(1):E271-5; discussion E276. doi: 10.1227/NEU.0b013e3181fe6165. PMID 21099705